CLINICAL TRIAL: NCT03450018
Title: An Open-label, Multi-center, Phase 1b Study to Investigate the Safety and Tolerability of SLC-0111 (WBI-5111) in Combination With Gemcitabine in Metastatic Pancreatic Ductal Adenocarcinoma Subjects Positive for Carbonic Anhydrase IX
Brief Title: A Study of SLC-0111 and Gemcitabine for Metastatic Pancreatic Ductal Cancer in Subjects Positive for CAIX
Acronym: SLC-0111-17-01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Changing treatment landscape: The availability of nab-paclitaxel with gemcitabine in the second-line setting has changed the feasibility of further recruitment and potential long-term development opportunities of SLC-0111 with gemcitabine alone.
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); SignalChem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-02841
Record Dates: First submitted 2018-02-13; First posted 2018-03-01 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Gemcitabine; SLC-0111; PDAC
MeSH Terms: interventions — SLC-0111; Gemcitabine

STUDY DESIGN:
Intervention Model Description: This is a traditional Phase I "3+3" study designed to identify the MTD by assessment of DLT of SLC-0111. Sample size estimates are not statistically based, but are based on acquisition of appropriate numbers of subjects to adequately describe the safety, tolerability, PK, and PD of SLC-0111 in combination with gemcitabine.
  Up to 18 subjects are anticipated to be enrolled in the dose escalation part; however, the actual number recruited will be dependent upon the number of dose escalations. Dose expansion (Part 2) may enroll up to 12 subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SLC-0111 + Gemcitabine (Experimental): Dose Level 1 - SLC-0111 (500 mg/day PO daily for 28 days) and Gemcitabine (1000 mg/m^2 IV on day 1, 8, and 15)
  Dose Level 2 - SLC-0111 (750 mg/day PO daily for 28 days) and Gemcitabine (1000 mg/m^2 IV on day 1, 8, and 15)
  Dose Level 3 - SLC-0111 (1000 mg/day PO daily for 28 days) and Gemcitabine (1000 mg/m^2 IV on day 1, 8, and 15)
  Interventions: Drug: SLC-0111; Drug: Gemcitabine Injection

INTERVENTIONS:
Drug: SLC-0111 — Oral SLC-0111
  Other Names: WBI-5111
Drug: Gemcitabine Injection — 1000 mg/m^2 IV
  Other Names: Gemcitabine

SUMMARY:
This is a multi-center, open-label Phase 1b study of SLC-0111 (oral) in combination with IV gemcitabine in CA IX positive subjects with mPDAC and comprises of 2 parts:

* Part 1: Dose Escalation
* Part 2: Dose Expansion

DETAILED DESCRIPTION:
This is a multi-center, open-label Phase 1b study of SLC-0111 (oral) in combination with IV gemcitabine in CA IX positive subjects with mPDAC and comprises of 2 parts:

* Part 1: Dose Escalation
* Part 2: Dose Expansion

Biopsy or archival tissue will be collected and tested for the presence of CAIX via Immunohistochemistry (IHC) and only subjects positive for CAIX will be enrolled in the dose-escalation and dose-expansion parts. Part 2 can only begin after a dosing regimen has been characterized in Part 1. Subjects who participated in Part 1 of study will not be eligible to participate in Part 2.

The dose escalation will aim to identify the safety, tolerability and MTD of the oral formulation of SLC-0111 in combination with IV gemcitabine. Additional subjects may be enrolled at the MTD in dose expansion cohort. Data collected will allow evaluation of safety, tolerability, PK, Pharmacodynamics (PD) and tumour response of SLC-0111 in combination with gemcitabine.

A traditional 3 + 3 dose escalation design will be utilized for this study. Cohorts (same dose level) of 3 to 6 evaluable subjects will participate in a dose escalation scheme in which the dose of SLC-0111 will be increased in each consecutive cohort. Dose escalation to a new cohort of subjects will occur after review of available Cycle 1 data. The dose of SLC-0111 will be escalated based on Table 1 and Table 2 in the protocol. Based on emerging data alternative dosing schedules, or dose reductions may be considered. Gemcitabine will be administered at the standard dose (1000 mg/m^2) and schedule (day 1, 8, and 15 of each cycle) but dose reductions may be considered if necessary.

* Each cohort will initially consist of up to 3 subjects.
* If none of the first 3 subjects in a cohort demonstrates dose limiting toxicities (DLTs), then the cohort will be declared safe and the next cohort will be opened for enrollment
* If 1 of the first 3 subjects in a cohort demonstrates DLTs, then 3 additional subjects will be accrued to that cohort for a total of 6 subjects
* If 1 out of 6 subjects in a cohort demonstrates DLTs, then the cohort will be declared safe and the next cohort (n=3)will be opened for enrollment
* If 2 or more subjects in a cohort demonstrates DLTs, that cohort will be declared to exceed the MTD

Following the identification of a Cohort that exceeds the MTD, the next lowest dose, or an intermediate dose level may be further explored.

The MTD will be defined as the highest dose level at which no more than 1 of 6 subjects demonstrates DLTs.

Intra-subject dose escalation will not be allowed in this study.

ELIGIBILITY:
Pre-Screening Inclusion Criteria:

* Males or females aged ≥ 18 years old.
* Able and willing to provide written pre-screening informed consent and to comply with the study protocol and procedures.
* A biopsiable tumour and a willingness to provide biopsies if no archival tumour tissue exists.
* Histologically or cytologically-confirmed metastatic pancreatic ductal adenocarcinoma (this can include distant lymph nodes). Subjects with locally advanced disease or regional lymph node involvement are to be excluded.

  * Regional lymph nodes are considered: Lymph nodes superior and inferior to head and body of pancreas, anterior and posterior pancreaticoduodenal, pyloric, proximal mesenteric nodes, and common bile duct lymph nodes, splenic hilar, pancreatic tail, peripancreatic, hepatic artery, infrapyloric (head only), subpyloric (head only), celiac (head only), superior mesenteric, pancreaticolienal (body and tail only), splenic (body and tail only), retroperitoneal, lateral aortic.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Life expectancy greater than 3 months in the investigator's opinion.
* Subject (archival tissue or pre-treatment biopsy) must be positive for CAIX via IHC before screening assessments listed below begin (i.e. Study Inclusion and Exclusion Criteria)

Main Study Inclusion Criteria:

* Males or females aged ≥ 18 years old.
* Able and willing to provide written informed consent and to comply with the study protocol and procedures.
* Histologically or cytologically-confirmed metastatic pancreatic ductal adenocarcinoma (this can include distant lymph nodes). Subjects with locally advanced disease or regional lymph node involvement are to be excluded.

  * Regional lymph nodes are considered: Lymph nodes superior and inferior to head and body of pancreas, anterior and posterior pancreaticoduodenal, pyloric, proximal mesenteric nodes, and common bile duct lymph nodes, splenic hilar, pancreatic tail, peripancreatic, hepatic artery, infrapyloric (head only), subpyloric (head only), celiac (head only), superior mesenteric, pancreaticolienal (body and tail only), splenic (body and tail only), retroperitoneal, lateral aortic.
* ≥1 prior line of systemic therapy with a 14-day washout period or if investigational combination is being considered for first line of therapy, subject was not eligible for FOLFIRINOX or gemcitabine + nab-paclitaxel.
* Recovery to ≤ Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies.
* ECOG performance status 0 or 1.
* Life expectancy greater than 3 months in the Investigator's opinion.
* The following time must have elapsed between previous therapy for cancer or medical history event and first administration of SLC-0111 and gemcitabine:

  * At least 2 weeks since previous cancer-directed therapy (cytotoxic agents, targeted therapy including monoclonal antibody therapy, immunotherapy, hormonal therapy, and prior radiotherapy).
  * At least 2 weeks or five times the elimination half-life (whichever is shortest) of any investigational drug/biologic or combination product prior to first dose of study treatment.
  * At least 4 weeks since any major surgery
  * At least 12 weeks since any incidence of severe gastrointestinal bleeding.
* Adequate renal function:

  * Creatinine ≤ 1.5 times upper limit of normal (ULN) or calculated creatinine clearance (CrCl) using the Cockcroft Gault formula ≥ 60 mL/min, or measured CrCl ≥ 60 mL/min.
* Adequate hepatic function:

  * Serum total bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN (≤ 5 x ULN if liver lesions present [i.e. liver metastasis or primary tumour of the liver for HCC]).
* Adequate hematologic function (without G-CSF support):

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Hemoglobin ≥ 85 g/L
* Adequate coagulation tests:

  * INR ≤ 1.5
  * PTT ≤ 1.5 times ULN
* Corrected QT interval (QTc) < 470 ms
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption.
* Negative pregnancy test in female subjects of child-bearing potential (defined as women who have not undergone hysterectomy/oophorectomy or who have not been naturally post-menopausal for ≥ 12 months).
* Subjects must agree not to donate gametes (oocyte or sperm) during study and for 4 months following last dose of study treatment.
* Sexually active subjects (male and female) must agree to use acceptable methods of contraception to avoid pregnancy prior to start of dosing, during the course of the study and for 4 months after the last dose of study treatment.
* Collect post-treatment biopsy if the tumour is biopsiable and a willingness to provide biopsies exists (optional)

Additional Inclusion Criteria for Dose Expansion (Part 2):

* Measurable disease as per RECIST 1.1.

Exclusion Criteria:

* Subjects negative for CAIX via IHC (biopsy or archival tissue)
* Previous treatment with any known CAIX Inhibitor
* Females who are pregnant, planning to become pregnant or breastfeeding.
* Severe cardiac disease which has required hospitalization within the past 3 months or which functionally limits a patient.
* Severe respiratory illness requiring supplemental oxygen or that significantly impacts functional status in daily life.
* Untreated CNS metastasis or CNS metastasis that has not been clinically stable for 28 days.
* History of myocardial infarction, unstable angina, congestive heart failure (New York Heart Association class ≥ III/IV), cerebrovascular accident, transient ischaemic attack, limb claudication at rest in the 6 months prior to enrolment, or ongoing symptomatic dysrhythmias, or uncontrolled atrial or ventricular arrhythmias, or uncontrolled hypertension.
* Any condition or illness that, in the opinion of the Investigator would compromise subject safety or interfere with the evaluation of the safety of the investigational products.
* Subjects with documented cases of human immunodeficiency virus (HIV) and viral load detectable.
* Hypersensitivity to investigational products or their excipients or severe allergy to sulfonamides.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, gastrointestinal bleeding, ulceration, or perforation within 12 weeks prior to the first administration of investigational products or significant bowel resection that would preclude adequate absorption.
* Known acute hepatitis B infection or chronic hepatitis B not currently on suppressive therapy.
* Known hepatitis C antibody positive and RNA positive. Subjects with hepatitis C antibody positivity but RNA negativity may enroll after consultation with hepatology.
* Active uncontrolled bacterial, viral, or fungal infections.
* Malignancy within the preceding 5 years (Subjects may be included in the trial if malignancy was a non-melanoma skin cancer, ductal carcinoma in-situ, early cervical malignancy, or at the discretion of the primary investigator if the malignancy has had curative intent treatment and has a < 10% chance of recurring within 5 years as per a well-recognized risk stratification tool specific for that malignancy.)

Additional Dose Expansion Exclusion Criteria:

Subjects cannot be enrolled in the dose expansion if they were enrolled during the dose escalation of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to Safety Follow-Up Visit (30 days +/- 7 days after permanently stopping study treatment)
  Adverse events (AEs) as assessed by CTCAE v5.0 will be determined by changes in safety assessments, including laboratory parameters, vital signs, ECG and physical examinations.

SECONDARY OUTCOMES:
The maximum tolerated dose [MTD] of SLC-0111 in combination with gemcitabine | Up to Safety Follow-Up Visit (30 days +/- 7 days after permanently stopping study treatment)
  Dose limiting toxicities (adverse events) will be determined by changes in safety assessments, including vital signs, clinical laboratory evaluations and ECG.
Maximum Plasma Concentration [Cmax] | Up to 4 years
  Analyze the pharmacokinetic profile of SLC-0111 and gemcitabine when used in combination by measuring the maximum (peak) plasma concentration (Cmax).
Time to Reach Maximum Plasma Concentraiton [Tmax] | Up to 4 years
  Analyze the pharmacokinetic profile of SLC-0111 and gemcitabine when used in combination by the time to reach maximum (peak) plasma concentration following drug administration (Tmax).
Elimination Rate Constant from the Central Compartment [Kel] | Up to 4 years
  Analyze the pharmacokinetic profile of SLC-0111 and gemcitabine when used in combination by measuring the elimination rate constant from the central compartment (Kel).
Volume of Distribution During Terminal Phase after Intravenous Administration [Vz] | Up to 4 years
  Analyze the pharmacokinetic profile of SLC-0111 and gemcitabine when used in combination by measuring the volume of distribution during terminal phase after intravenous administration (Vz).
Area Under the Concentration-Time Curve from Zero up to a Definite Time T [AUC(0-T)] | Up to 4 years
  Analyze the pharmacokinetic profile of SLC-0111 and gemcitabine when used in combination by measuring the area under the concentration-time curve from zero up to a definite time T (AUC(0-T)).
Area Under the Concentration-Time Curve from Zero up to Infinity [AUC(0-inf)] | Up to 4 years
  Analyze the pharmacokinetic profile of SLC-0111 and gemcitabine when used in combination by measuring the area under the concentration-time curve from zero up to infinity with extrapolation of the terminal phase (AUC(0-inf)).
Elimination Half-Life | Up to 4 years
  Analyze the pharmacokinetic profile of SLC-0111 and gemcitabine when used in combination by measuring the elimination half-life (T1/2).
Determine the Recommended Phase II Dose of SLC-0111 in combination with gemcitabine | Up to 2 years
  Recommended Phase II Dose (RP2D) Safety and PK
Objective Response Rate [ORR] as Assessed by RECIST 1.1 | Up to 1 year
  Objective response rate (ORR) as assessed by RECIST 1.1 or clinical examination, where appropriate. ORR is the change in tumour volume from baseline to best overall response.
Progression-Free Survival [PFS] as Assessed by RECIST 1.1 | Up to 1 year
  Progression-free survival (PFS) as assessed by RECIST 1.1 or clinical examination, where appropriate. PFS is defined as the duration of time from start of treatment to progression or death, whichever occurs first. Subjects alive at the time of last follow up without disease progression will be censored at that time point.
Duration of Response as Assessed by RECIST 1.1 | Up to 2 years
  Duration of response as assessed by RECIST 1.1 or clinical examination, where appropriate. Duration of response is defined as the time from start of response [Complete Response (CR) or Partial Response (PR)] until progression or death due to any cause.
Overall Survival [OS] | Up to the end of the study
  Overall survival (OS) is defined as the time from initiation of investigational product(s) to death due to any cause.

OTHER OUTCOMES:
Tumour Metabolic Response Using Positron Emission Tomography with 18F-FDG-PET | Up to C3D1 +/- 7 days
  Changes in mean standard values of 18F-FDG uptake expressed as the peak standardized uptake value corrected for lean body mass (SULpeak),as defined by Positron Emission Tomography (PET) Response Criteria in Solid Tumours (PERCIST 1.0)
CAIX Biomarker Values | Up to 4 years
  Change from baseline in CAIX biomarker measured in tumour biopsies. Explore relationships between CAIX biomarker values and markers of clinical activity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Renouf, MD, Principal Investigator — BC Cancer - Vancouver
Locations (2):
- Canada (2):
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Assaf E, Verlinde-Carvalho M, Delbaldo C, Grenier J, Sellam Z, Pouessel D, Bouaita L, Baumgaertner I, Sobhani I, Tayar C, Paul M, Culine S. 5-fluorouracil/leucovorin combined with irinotecan and oxaliplatin (FOLFIRINOX) as second-line chemotherapy in patients with metastatic pancreatic adenocarcinoma. Oncology. 2011;80(5-6):301-6. doi: 10.1159/000329803. Epub 2011 Jul 18. PMID 21778770
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Chang Q, Jurisica I, Do T, Hedley DW. Hypoxia predicts aggressive growth and spontaneous metastasis formation from orthotopically grown primary xenografts of human pancreatic cancer. Cancer Res. 2011 Apr 15;71(8):3110-20. doi: 10.1158/0008-5472.CAN-10-4049. Epub 2011 Feb 22. PMID 21343390
- [Background] Choi SW, Kim JY, Park JY, Cha IH, Kim J, Lee S. Expression of carbonic anhydrase IX is associated with postoperative recurrence and poor prognosis in surgically treated oral squamous cell carcinoma. Hum Pathol. 2008 Sep;39(9):1317-22. doi: 10.1016/j.humpath.2007.10.026. Epub 2008 Apr 28. PMID 18440050
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Couvelard A, O'Toole D, Leek R, Turley H, Sauvanet A, Degott C, Ruszniewski P, Belghiti J, Harris AL, Gatter K, Pezzella F. Expression of hypoxia-inducible factors is correlated with the presence of a fibrotic focus and angiogenesis in pancreatic ductal adenocarcinomas. Histopathology. 2005 Jun;46(6):668-76. doi: 10.1111/j.1365-2559.2005.02160.x. PMID 15910598
- [Background] Coveler AL, Herman JM, Simeone DM, Chiorean EG. Localized Pancreatic Cancer: Multidisciplinary Management. Am Soc Clin Oncol Educ Book. 2016;35:e217-26. doi: 10.1200/EDBK_160827. PMID 27249726
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Erkan M, Kurtoglu M, Kleeff J. The role of hypoxia in pancreatic cancer: a potential therapeutic target? Expert Rev Gastroenterol Hepatol. 2016;10(3):301-16. doi: 10.1586/17474124.2016.1117386. Epub 2015 Nov 27. PMID 26560854
- [Background] Gieling RG, Parker CA, De Costa LA, Robertson N, Harris AL, Stratford IJ, Williams KJ. Inhibition of carbonic anhydrase activity modifies the toxicity of doxorubicin and melphalan in tumour cells in vitro. J Enzyme Inhib Med Chem. 2013 Apr;28(2):360-9. doi: 10.3109/14756366.2012.736979. Epub 2012 Nov 19. PMID 23163664
- [Background] Guillaumond F, Leca J, Olivares O, Lavaut MN, Vidal N, Berthezene P, Dusetti NJ, Loncle C, Calvo E, Turrini O, Iovanna JL, Tomasini R, Vasseur S. Strengthened glycolysis under hypoxia supports tumor symbiosis and hexosamine biosynthesis in pancreatic adenocarcinoma. Proc Natl Acad Sci U S A. 2013 Mar 5;110(10):3919-24. doi: 10.1073/pnas.1219555110. Epub 2013 Feb 13. PMID 23407165
- [Background] Kon-no H, Ishii G, Nagai K, Yoshida J, Nishimura M, Nara M, Fujii T, Murata Y, Miyamoto H, Ochiai A. Carbonic anhydrase IX expression is associated with tumor progression and a poor prognosis of lung adenocarcinoma. Lung Cancer. 2006 Dec;54(3):409-18. doi: 10.1016/j.lungcan.2006.08.017. Epub 2006 Oct 9. PMID 17030461
- [Background] Koong AC, Mehta VK, Le QT, Fisher GA, Terris DJ, Brown JM, Bastidas AJ, Vierra M. Pancreatic tumors show high levels of hypoxia. Int J Radiat Oncol Biol Phys. 2000 Nov 1;48(4):919-22. doi: 10.1016/s0360-3016(00)00803-8. PMID 11072146
- [Background] McDonald PC, Winum JY, Supuran CT, Dedhar S. Recent developments in targeting carbonic anhydrase IX for cancer therapeutics. Oncotarget. 2012 Jan;3(1):84-97. doi: 10.18632/oncotarget.422. PMID 22289741
- [Background] O JH, Lodge MA, Wahl RL. Practical PERCIST: A Simplified Guide to PET Response Criteria in Solid Tumors 1.0. Radiology. 2016 Aug;280(2):576-84. doi: 10.1148/radiol.2016142043. Epub 2016 Feb 24. PMID 26909647
- [Background] Oettle H, Neuhaus P, Hochhaus A, Hartmann JT, Gellert K, Ridwelski K, Niedergethmann M, Zulke C, Fahlke J, Arning MB, Sinn M, Hinke A, Riess H. Adjuvant chemotherapy with gemcitabine and long-term outcomes among patients with resected pancreatic cancer: the CONKO-001 randomized trial. JAMA. 2013 Oct 9;310(14):1473-81. doi: 10.1001/jama.2013.279201. PMID 24104372
- [Background] Pacchiano F, Carta F, McDonald PC, Lou Y, Vullo D, Scozzafava A, Dedhar S, Supuran CT. Ureido-substituted benzenesulfonamides potently inhibit carbonic anhydrase IX and show antimetastatic activity in a model of breast cancer metastasis. J Med Chem. 2011 Mar 24;54(6):1896-902. doi: 10.1021/jm101541x. Epub 2011 Mar 1. PMID 21361354
- [Background] Portal A, Pernot S, Tougeron D, Arbaud C, Bidault AT, de la Fouchardiere C, Hammel P, Lecomte T, Dreanic J, Coriat R, Bachet JB, Dubreuil O, Marthey L, Dahan L, Tchoundjeu B, Locher C, Lepere C, Bonnetain F, Taieb J. Nab-paclitaxel plus gemcitabine for metastatic pancreatic adenocarcinoma after Folfirinox failure: an AGEO prospective multicentre cohort. Br J Cancer. 2015 Sep 29;113(7):989-95. doi: 10.1038/bjc.2015.328. Epub 2015 Sep 15. PMID 26372701
- [Background] Sirri E, Castro FA, Kieschke J, Jansen L, Emrich K, Gondos A, Holleczek B, Katalinic A, Urbschat I, Vohmann C, Brenner H. Recent Trends in Survival of Patients With Pancreatic Cancer in Germany and the United States. Pancreas. 2016 Jul;45(6):908-14. doi: 10.1097/MPA.0000000000000588. PMID 26745860
- [Background] Sohal DP, Mangu PB, Laheru D. Metastatic Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline Summary. J Oncol Pract. 2017 Apr;13(4):261-264. doi: 10.1200/JOP.2016.017368. Epub 2016 Oct 31. No abstract available. PMID 28399388
- [Background] Supuran CT. Carbonic anhydrases: novel therapeutic applications for inhibitors and activators. Nat Rev Drug Discov. 2008 Feb;7(2):168-81. doi: 10.1038/nrd2467. PMID 18167490
- [Background] Supuran CT. Drug interaction considerations in the therapeutic use of carbonic anhydrase inhibitors. Expert Opin Drug Metab Toxicol. 2016;12(4):423-31. doi: 10.1517/17425255.2016.1154534. Epub 2016 Mar 3. PMID 26878088
- [Background] Supuran CT. How many carbonic anhydrase inhibition mechanisms exist? J Enzyme Inhib Med Chem. 2016;31(3):345-60. doi: 10.3109/14756366.2015.1122001. Epub 2015 Nov 30. PMID 26619898
- [Background] Tsai S, Evans DB. Therapeutic Advances in Localized Pancreatic Cancer. JAMA Surg. 2016 Sep 1;151(9):862-8. doi: 10.1001/jamasurg.2016.1113. PMID 27276001
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Background] Zhang Y, Hochster H, Stein S, Lacy J. Gemcitabine plus nab-paclitaxel for advanced pancreatic cancer after first-line FOLFIRINOX: single institution retrospective review of efficacy and toxicity. Exp Hematol Oncol. 2015 Oct 7;4:29. doi: 10.1186/s40164-015-0025-y. eCollection 2015. PMID 26451276